CLINICAL TRIAL: NCT06183008
Title: Effect of Intravenous Immunoglobulins on Painful Sensory Neuropathy Evaluated by Aggregated N-of-one Trials
Brief Title: IVIG in Painful Sensory Neuropathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other); University Hospital of North Norway (Other); University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVIGSeN
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-03

CONDITIONS: Sensory Neuropathy; Small Fiber Neuropathy
Keywords: nervous system diseases; neuromuscular diseases; peripheral nervous system diseases; small fiber neuropathy; sensory neuronopathy; sensory neuropathy; IVIG; Intravenous immunoglobulin; n-of-1; Sørlandet sykehus; Sorlandet hospital; Kristiansand; polyneuropathy; Intravenous immune globulin
MeSH Terms: conditions — Small Fiber Neuropathy; Nervous System Diseases; Neuromuscular Diseases; Peripheral Nervous System Diseases; Polyneuropathies | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Intervention Model Description: N-of-one trial, individual randomized, double-blind, and multiple crossover comparisons of an interventional treatment and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Immunoglobulin (Experimental): 3 courses Intravenous immunoglobulin, Infusion solution, 100mg/ml, 2g/kg over 3 days
  Interventions: Drug: Intravenous immunoglobulin
- Placebo (Placebo Comparator): 3 courses Saline infusion solution 0,9%, same volume as IVIG over 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous immunoglobulin — Each patient will during the 30-week trial period get 3 IVIG courses (each total dose 2g/kg) for three consecutive days
  Other Names: IVIG; Privigen
  Arms: Intravenous Immunoglobulin
Drug: Placebo — Each patient will during the 30-week trial period get 3 placebo courses (each 0.9% saline similar volume) for three consecutive days
  Other Names: 0.9% saline
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess effect of Intravenous immunoglobulins (antibodies) as compared to Placebo, on pain intensity in patients from 18-65 years with painful sensory neuropathy without a known cause. Effect of the treatment will be recorded by the patient in a digital diary.

DETAILED DESCRIPTION:
Patients suffering from idiopathic sensory neuropathies often report excruciating pain that interferes with daily function and leads to impaired quality of life. Current neuropathic pain treatment options are in general insufficient. Autoimmunity may play a role in some patients, and treatment with intravenous immunoglobulins (IVIG) may have a potential beneficial effect. Available scientific documentation on this topic is limited and disparate.

The main purpose of this trial is to assess effect of IVIG as compared to placebo on pain intensity in patients >18 years with idiopathic painful small fiber neuropathy or sensory neuronopathy.

Each patient will during the 30-week trial period get 3 IVIG courses and 3 placebo courses in a randomized order, given every 5 week on an outpatient basis for three consecutive days. Outcome measures will be recorded by the patient in a digital diary

ELIGIBILITY:
Inclusion Criteria:

Painful sensory neuropathy fulfilling diagnostic criteria for idiopathic small fiber neuropathy or sensory neuronopathy

* Idiopathic small fiber neuropathy (all of the following)

  1. Neuropathic pain (length-dependent/non-length dependent/focal) and at least two of the following clinical signs

     1. Hypoesthesia (tactile, pinprick, or thermal)
     2. Allodynia (tactile, dynamic, thermal, pressure)
     3. Hyperalgesia
     4. Aftersensation
  2. Normal nerve conduction studies:
  3. Reduced intra-epidermal nerve fiber density at the distal leg (IENFD) at the distal leg or Reduced thermal threshold assessed at the foot by QST
  4. Causal investigation according to clinical guidelines has not revealed a cause of the neuropathy
* Sensory neuronopathy (all of the following)

  1. Clinical pure sensory neuropathy
  2. A score >6.5 on the following

     1. Ataxia in the lower or upper limb: 3.1p
     2. Asymmetrical distribution of sensory loss: 1.7p IVIGSeN Protocol number 1.2
     3. Sensory loss not restricted to the lower limb at full development: 2.0 p
     4. At least 1 sensory action potential absent or 3 sensory action potentials <30% of the lower limit of normal in the upper limbs not explained by entrapment neuropathy: 2.8p
     5. Less than two nerves with abnormal motor nerve conduction studies in the lower limbs: 3.1p
  3. Causal investigation according to clinical guidelines has not revealed a cause of the neuropathy

Pain intensity > 5.0 on a pain score from 0-10, lasting at least 4 weeks

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Previous allergic reaction to IVIG or other blood products)
2. Selective IgA deficiency
3. Cardiac insufficiency (NYHA III/IV ie marked or severe limitation in activity due to symptoms, even during less-than-ordinary activity)
4. Cardiac dysrhythmia requiring treatment
5. Unstable or advanced ischemic heart disease
6. Severe hypertension (diastolic >120 or systolic > 170)
7. Known hyperviscosity
8. Renal insufficiency (GFR < 30 ml/min/1,73m2) or nephrotic syndrome
9. Previous thromboembolic event
10. Smoking
11. Diabetes
12. Prolonged immobilization
13. Hypercoagulable state

    Prior/Concomitant Therapy
14. Change of pain medication in the 30 days prior to inclusion (unchanged pain medication is allowed, provided dosages stay equal during the study)
15. Treatment with IVIG the last 4 weeks or other ongoing immunomodulatory treatments
16. Use of loop diuretics, Dinutuksimab beta, or Imlifidase Diagnostic assessments
17. Predominant clinical or neurographic features of motor nerve fiber involvement Other Exclusions
18. Females who are breastfeeding, pregnant or unwilling to practice contraception throughout the study
19. Unable to give independent informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity the second week | The second week after start of IVIG/Placebo infusions (mean of days 8, 10 and 13)
  Pain intensity after IVIG/Placebo infusions scored on a numeric rating scale (NRS) ranging from 0 to 10

SECONDARY OUTCOMES:
Pain intensity across 4 weeks | Day 8 to 34 after start of each infusion
  Pain intensity across 4 weeks after start of each infusion (mean of scoring three times per week from)
Disability and quality of life | At the end of the third week after infusion
  Scored on: Polyneuropathy Patient-reported Index (CAPPRI)
Anti-FGF3 antibodies | Before start of infusion of IVIG/Placebo week 1, 5, 11, 16, 21 and 26
  Blood samples will be tested for anti-FGF3 antibodies to evaluate their association with the observed clinical response in terms of pain relief to IVIG.
Adverse events | From start to end of interventions week 1 - 30
  Recording adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Marius Ørnes, Cand.med, Principal Investigator — Sorlandet Hospital HF, Department of Neurology; Unn Ljøstad, Cand.med PhD, Study Director — Sorlandet Hospital HF, Department of Neurology; Åse Mygland, Cand.med PhD, Study Director — Sorlandet Hospital HF, Department of Neurology